CLINICAL TRIAL: NCT04780061
Title: Dietary Supplements to Reduce Symptom Severity and Duration in People With SARS-CoV-2: A Randomized, Double Blind, Placebo Controlled Clinical Trial
Brief Title: Dietary Supplements for COVID-19
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Public PCR testing stopped in Ontario
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: Ottawa Hospital Research Institute (Other); Vitazan Professional (Other); New Roots Herbal (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20210072-01H
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Covid19
Keywords: Natural Health Products; NHP; Dietary Supplements; Vitamin C; Vitamin D; Vitamin K; Zinc; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Cholecalciferol; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Specific Product: Vitamin D3 50,000 IU
  Formulation: Capsule. Each capsule will contain 500 mg (50,000 units) cholecalciferol (vitamin D3) Dose: One capsule on day 1 of the intervention period
  Specific Product: Vitamin K2/D
  Formulation: Liquid. Each 0.0285 mL drop contains 30 mcg menaquinone-7 (MK-7, vitamin K2) and 3.125 mcg (125 units) cholecalciferol (vitamin D3).
  Dose: 0.114 mL (four drops) twice daily for 21 days totalling 240mcg MK-7 and 1,000 units cholecalciferol per day.
  Specific Product: Vitamin C/Zinc
  Formulation: Capsule. Each capsule will contain 666 mg ascorbic acid (vitamin C) and 8.3 mg of zinc acetate Dose: Three capsules three times daily for 21 days totalling 6 g ascorbic acid and 75 mg zinc acetate per day.
  Interventions: Drug: Vitamin D3 50,000 IU; Dietary Supplement: Vitamin C/Zinc; Dietary Supplement: Vitamin K2/D
- Control (Placebo Comparator): Specific Product: Vitamin D3 50,000 IU
  Placebo Equivalent: microcrystalline cellulose capsule, 350 mg
  Specific Product: Vitamin K2/D
  Placebo Equivalent: Medium chain triglyceride oil
  Specific Product: Vitamin C/Zinc
  Placebo Equivalent: microcrystalline cellulose capsule, 350 mg
  Interventions: Other: Microcrystalline Cellulose Capsule; Other: Medium Chain Triglyceride Oil

INTERVENTIONS:
Drug: Vitamin D3 50,000 IU — This is a loading dose of Vitamin D. Vitamin D (cholecalciferol [vitamin D3]) is a fat-soluble vitamin that is synthesized following ultraviolet radiation to the skin, naturally occurs in a few dietary sources and is available as a dietary supplement.
  Other Names: Cholecalciferol
  Arms: Treatment
Dietary Supplement: Vitamin C/Zinc — This is a combination of Vitamin C and Zinc. Vitamin C (ascorbic acid, ascorbate) is a water-soluble vitamin that naturally occurs in many foods and is sold as a dietary supplement. It is required for the functioning of several enzymes and is important for the immune system. Zinc is one of the most abundant essential trace elements in the human body and is required for the function of several hundred enzymes and transcription factors.
  Arms: Treatment
Dietary Supplement: Vitamin K2/D — This is a combination of Vitamin K2 (menaquinone-7) and vitamin D. Vitamin K (menaquinone-7 [vitamin K2]) is a fat-soluble vitamin found in foods and sold as a dietary supplement. Vitamin K plays a large role in synthesizing coagulation factors in the blood, and vitamin K deficiency has been associated with uncontrolled bleeding. Vitamin K1 (phylloquinone) is an alternate form of vitamin K found in foods and supplements; however, vitamin K2 has a better absorption profile50 and additionally plays a role in bone metabolism controlling the binding of calcium, especially in older adults, where it attenuates the rate of bone loss
  Arms: Treatment
Other: Microcrystalline Cellulose Capsule — Placebo equivalent of Vitamin C/Zinc and Vitamin D3.
  Arms: Control
Other: Medium Chain Triglyceride Oil — Placebo equivalent of Vitamin K2/D
  Arms: Control

SUMMARY:
This is a double blind, placebo controlled, phase III randomized controlled trial evaluating the effects of the dietary supplements vitamin C, vitamin D, vitamin K, and zinc versus placebo on the overall health, symptom severity, and symptom duration of outpatients diagnosed with SARS-CoV-2.

DETAILED DESCRIPTION:
This study proposed is a double-blind, placebo-controlled, phase III randomized controlled trial powered to detect meaningful differences in the overall health and symptom severity of people with COVID-19 between the treatment and control arms. Eligible participants will be randomly assigned, using a web randomization system, in a ratio of 1:1 to one of the following groups: (1) nutrient therapy with vitamin D, vitamin C, vitamin K2, and zinc or (2) placebo. Total trial duration will be 12 weeks. Nutrients or placebo will be given for a period of 21 days following enrolment and randomization. Total trial duration will be 12 weeks. Adverse events will be collected during the treatment phase plus one additional week (maximum 4 weeks).

With respect to the primary outcome of participant-reported overall health, power calculations were conducted based on between-group differences at a single time point (21 days) and Cohen's guideline for a small effect size of 0.3. A sample size of 176 (88 per arm) provides 80% power to detect a difference at an α of 0.05. To account for an approximate 10-15% lost to follow-up we will enrol 200 participants (100 per arm).

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18) who test positive for SARS-CoV-2 in an outpatient setting
2. Access to internet

Exclusion Criteria:

1. Symptom onset greater than 4 days prior to enrolment
2. Supplementing regularly with >500 mg vitamin C, >1000 units vitamin D, >120 mcg vitamin K (any form), or >15 mg zinc taken daily within the past month
3. Currently taking warfarin or an equivalent vitamin K antagonist anticoagulant
4. End stage chronic kidney disease
5. History of calcium oxalate kidney stones
6. Active granulomatosis (sarcoidosis, tuberculosis, lymphoma)
7. Known hypercalcemia or hypervitaminosis D
8. Currently taking either of the following antibiotics: cephalexin, tetracyclines
9. Participating in an investigational study or participation in an investigational study within the past 30 days
10. Any reason which, under the discretion of the qualified investigator or delegate, would preclude the patient from participating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dugald Seely, ND, MSc, Principal Investigator — Canadian College of Naturopathic Medicine; Kumanan Wilson, MD, MSc, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Centre for Health Innovation, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seely D, Legacy M, Conte E, Keates C, Psihogios A, Ramsay T, Fergusson DA, Kanji S, Simmons JG, Wilson K. Dietary supplements to reduce symptom severity and duration in people with SARS-CoV-2: a double-blind randomised controlled trial. BMJ Open. 2023 Sep 22;13(9):e073761. doi: 10.1136/bmjopen-2023-073761. PMID 37739466
- [Derived] Legacy M, Seely D, Conte E, Psihogios A, Ramsay T, Fergusson DA, Kanji S, Simmons JG, Wilson K. Dietary supplements to reduce symptom severity and duration in people with SARS-CoV-2: study protocol for a randomised, double-blind, placebo controlled clinical trial. BMJ Open. 2022 Mar 3;12(3):e057024. doi: 10.1136/bmjopen-2021-057024. PMID 35241474

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from outpatient COVID-19 test centres associated with The Ottawa Hospital. The primary site for enrolment and coordination of the study was The Centre for Health Innovation, Ottawa, Canada with support from the Ottawa Hospital Research Institute.
Groups:
- Treatment: Vitamin C 6g Oral Daily x 21 Days; Vitamin D3 50,000 IU Oral x1; Vitamin D3 1,000 IU Oral Daily x 21 Days; Vitamin K2 240 mcg Oral Daily x 21 Days; Zinc Acetate 75mg Oral Daily x 21 Days;
- Control: Placebo (Microcrystalline cellulose + medium chain triglyceride oil). Number of pills, frequency, and duration identical to treatment arm.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 44 | 46
Treated | 42 (Two participants started study but were withdrawn before they began treatment) | 44 (Two participants started study but were withdrawn before they began treatment)
Completed | 36 | 31
Not Completed | 8 | 15
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Population: Participants only included if they began study treatments.
Groups:
- Treatment: Vitamin C, Vitamin D3, Vitamin K2, Zinc
- Control: Placebo (Microcrystalline cellulose + medium chain triglyceride oil)
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (12.7) | 39.9 (14.9) | 38.9 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 26 | 43
  Male | 25 | 18 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race data missing for 4 participants in the control arm
  Participants
    Black: number analyzed (Participants) | 42 | 40 | 82
    Black | 1 | 2 | 3
    White: number analyzed (Participants) | 42 | 40 | 82
    White | 37 | 34 | 71
    Latin American: number analyzed (Participants) | 42 | 40 | 82
    Latin American | 1 | 0 | 1
    Asian (South): number analyzed (Participants) | 42 | 40 | 82
    Asian (South) | 0 | 1 | 1
    Asian (Southeast): number analyzed (Participants) | 42 | 40 | 82
    Asian (Southeast) | 1 | 1 | 2
    Asian (East): number analyzed (Participants) | 42 | 40 | 82
    Asian (East) | 0 | 2 | 2
    Middle Eastern: number analyzed (Participants) | 42 | 40 | 82
    Middle Eastern | 2 | 0 | 2
Vaccination Status [Count of Participants; unit: Participants]
  Received First Dose | 41 | 42 | 83
  Received Second Dose | 41 | 42 | 83
  Received Third Dose | 37 | 30 | 67
  Unvaccinated | 1 | 2 | 3
Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 3 | 1 | 4
  Diabetes | 0 | 2 | 2
  Coronary Artery Disease | 0 | 0 | 0
  Asthma | 7 | 9 | 16
  Chronic Kidney Disease | 0 | 0 | 0
  Chronic Obstructive Pulmonary Disorder | 0 | 2 | 2
  Liver Disease | 0 | 0 | 0
  Cancer | 0 | 1 | 1
  Immunodeficiency | 0 | 0 | 0
Other Variables [Count of Participants; unit: Participants]
  Smoking History | 7 | 8 | 15
  Symptoms at Testing | 38 | 36 | 74

OUTCOME MEASURES:

1. Primary Outcome: Participant-reported Overall Health
Description: Measured using the EuroQol Visual Assessment Scale (EQ-VAS). Scores each day range from 0 (worst health imaginable) and 100 (best health imaginable). Scores summed over a 21-day period for a total range of 0-2100.
Time Frame: During the intervention period (Daily for 21 days)
Population: Participants were included in the analysis of overall health, symptom severity, and symptom duration if they completed the 21-day intervention period, completed at least 11 (52%) daily assessments, and did not miss more than 3 assessments sequentially
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 34 | 24
score on a scale | 1790 (226.6) | 1752.6 (220.7)
Statistical Analysis 1: Comparison: Treatment vs Control; An area under the curve approach was used to analyze the primary outcome, whereby participants' scores for each assessment were summed over the 21-day period. For missing values, we imputed the mean of the most recent and first subsequent measurement or carried the last observation forward if there was no subsequent measurement; Test type: Superiority; p = 0.53, t-test, 2 sided

2. Secondary Outcome: Effect of COVID-19 on the Health Status of Participants
Description: Measured using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire. Scores are converted into a unique health state. Health states are converted to an index value between 0 and 1, where 1 is considered the best possible health and 0 is the worst possible health.
Time Frame: Baseline plus weeks 1, 2, 3, 4, 8, and 12
Population: Participants were included in this analysis if they completed a baseline questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 41 | 40
score on a scale
  Baseline | 0.88 (0.1) | 0.88 (0.12)
  Week 1 | 0.95 (0.08) | 0.93 (0.1)
  Week 2 | 0.95 (0.07) | 0.94 (0.09)
  Week 3 | 0.94 (0.08) | 0.91 (0.1)
  Week 4 | 0.96 (0.08) | 0.97 (0.05)
  Week 8 | 0.95 (0.08) | 0.95 (0.09)
  Week 12 | 0.96 (0.07) | 0.96 (0.07)

3. Secondary Outcome: Symptom Severity of Common COVID-19 Symptoms
Description: Measured using an internally-developed questionnaire. Includes fever, cough, shortness of breath, fatigue, headache, myalgia/arthralgia, nausea, vomiting, diarrhea, congestion, loss of taste, and loss of smell. Scores range from 0-3 for each symptom, totaling 0-42 for each day. 0 = no symptom, 1 = mild symptom, 2 = moderate symptom, 3 = severe symptom. Scores converted into a number out of 100 and summed over 21 days for a range of 0-2100 where a higher score indicates a higher symptom severity (i.e., a worse outcome).
Time Frame: During the intervention period (Daily for 21 days)
Population: Participants were included in this analysis if they completed the 21-day intervention period, completed at least 11 (52%) daily assessments, and did not miss more than 3 assessments sequentially.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 34 | 24
score on a scale | 166.3 (92.3) | 192.9 (153.6)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.09, t-test, 2 sided

4. Secondary Outcome: Total Symptom Duration
Description: Measured as the time to a complete reduction of symptoms with no relapses (i.e., a 0 in all categories on the symptom questionnaire).
Time Frame: During the intervention period (21 days)
Population: as for outcome 3
Measure: Median (Full Range); unit: Days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 34 | 24
Days | 13.0 [0 to 21] | 12.5 [0 to 21]
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.81, Log Rank

5. Secondary Outcome: Incidence of Delayed Return to Usual Health
Description: Measured by the number of people experiencing "ongoing symptomatic COVID-19" (symptoms persisting between 4 and 12 weeks) and the number of people experiencing "post-COVID-19 syndrome" (symptoms persisting at least 12 weeks)
Time Frame: 12 weeks
Population: Participants were included in this analysis if they completed 12 weeks of follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 35 | 28
Participants
  Ongoing Symptomatic COVID-19 | 6 | 5
  Post COVID-19 Syndrome | 3 | 3

6. Secondary Outcome: Number of Participants With a Hospital Visit or Admission
Description: Includes ER visits, acute care admissions, and ICU admissions
Time Frame: 12 weeks
Population: All participants who started the study drug were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 42 | 44
Participants
  Emergency Room Visits | 2 | 4
  Acute Care Admissions | 0 | 0
  Intensive Care Unit Admissions | 0 | 0

ADVERSE EVENTS:
Time Frame: During the intervention period (21 days) plus 1 additional week (4 weeks total)
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/44 | 1/46
Other Adverse Events (participants affected / at risk) | 16/44 | 6/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=44) | Control (N=46)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=44) | Control (N=46)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
Jaw Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed; Symptom severity and duration questionnaire not validated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT04780061/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT04780061/ICF_001.pdf